CLINICAL TRIAL: NCT05523739
Title: A Randomized, Double-Blind, Placebo-Controlled, Phase I Clinical Study Evaluating the Safety of a Single Ascending Dose of STI-1558 in Healthy Subjects and the Safety, Pharmacokinetics, and Efficacy of Multiple Ascending Doses of STI-1558 in SARS-CoV-2-Positive Subjects
Brief Title: Safety and Efficacy Study of STI-1558 in Healthy Adults and SARS-CoV-2-Positive Patients
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Zhejiang ACEA Pharmaceutical Co. Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: MPR-COV-101CN
Record Dates: First submitted 2022-08-25; First posted 2022-08-31 (Actual); Last update posted 2023-08-14 (Actual); Status verified 2023-08

CONDITIONS: SARS-CoV-2 Infection
MeSH Terms: conditions — COVID-19 | interventions — STI-1558

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (7):
- Part 1: Cohort 1 (Experimental): Participants will receive a single 300 mg dose of STI-1558 or placebo. Cohort 1 will dose 6 subjects to STI-1558 and 2 subjects to placebo.
  Interventions: Drug: STI-1558
- Part 1: Cohort 2 (Experimental): Participants will receive a single 600 mg dose of STI-1558 or placebo. Cohort 2 will dose 6 subjects to STI-1558 and 2 subjects to placebo.
  Interventions: Drug: STI-1558
- Part 1: Cohort 3 (Experimental): Participants will receive a single 1200 mg dose of STI-1558 or placebo. Cohort 3 will dose 6 subjects to STI-1558 and 2 subjects to placebo.
  Interventions: Drug: STI-1558
- Part 1: Cohort 4 (Experimental): Participants will receive a single 2000 mg dose of STI-1558 or placebo. Cohort 4 will dose 6 subjects to STI-1558 and 2 subjects to placebo.
  Interventions: Drug: STI-1558
- Part 2: Cohort 1 (Experimental): Participants will receive a 300 mg dose of STI-1558 or placebo q12h on Day1 to Day7 and once in the morning on Day8 for a total of 15 doses.
  Cohort 1 will dose 6 subjects to STI-1558 and 2 subjects to placebo.
  Interventions: Drug: STI-1558
- Part 2: Cohort 2 (Experimental): Participants will receive a 600 mg dose of STI-1558 or placebo q12h on Day1 to Day7 and once in the morning on Day8 for a total of 15 doses.
  Cohort 2 will dose 16 subjects to STI-1558 and 8 subjects to placebo.
  Interventions: Drug: STI-1558
- Part 2: Cohort 3 (Experimental): Participants will receive a 800 mg dose of STI-1558 or placebo q12h on Day1 to Day7 and once in the morning on Day8 for a total of 15 doses.
  Cohort 3 will dose 16 subjects to STI-1558 and 8 subjects to placebo.
  Interventions: Drug: STI-1558

INTERVENTIONS:
Drug: STI-1558 — An oral small molecule prodrug that effectively inhibits the SARS-CoV-2 main protease (Mpro).

SUMMARY:
The purpose of this study is to evaluate the safety of STI-1558 in healthy subjects and the safety, pharmacokinetics, and efficacy in SARS-CoV-2-Positive subjects.

DETAILED DESCRIPTION:
This is a two-part, randomized, double-blind, placebo-controlled study evaluating the safety and pharmacokinetics (PK) of a single ascending dose of STI-1558 in healthy subjects and the safety, PK and efficacy of a multiple ascending dose in SARS-CoV-2-positive subjects.

ELIGIBILITY:
Inclusion Criteria:

* Part 1

  1. Subjects are fully informed of the study and sign the informed consent document prior to any procedure.
  2. Healthy subjects aged ≥18 but ≤45 years old, regardless of gender.
  3. BMI ≥18, but ≤30kg/m2, and weight ≥45, but ≤100kg.
  4. Good health status, with normal or abnormal and not clinically significant (NCS) results of medical history, vital signs, physical examination, 12-lead electrocardiogram, laboratory tests (blood routine, blood chemistry, urine routine, coagulation function) and thyroid function (TSH, FT3, FT4) during the screening period.
  5. Must be willing and able to comply with all planned study procedures.
  6. Women of childbearing potential (WOCBP) (infertile women defined as having undergone hysterectomy or bilateral oophorectomy or bilateral salpingectomy or bilateral tubal ligation/closure, or who are infertile due to a congenital or acquired condition or spontaneously menopausal for ≥ 12 months) must have a negative blood pregnancy test during screening. Fertility female and male subjects must use a highly effective method of contraception from the screening period to 90 days after the last dose of study drug.
* Part 2

  1. Subjects are fully informed of the study and sign the informed consent document prior to any procedure.
  2. Age ≥ 18, but < 65 years old, gregardless of gender.
  3. BMI ≥18, but ≤30kg/m2, and weight ≥45, but ≤100kg.
  4. Asymptomatic or mild patients diagnosed with SARS-CoV-2 positive according to the Diagnosis and Treatment Protocol for Novel Coronavirus Pneumonia (Trial Version 9).
  5. First positive for SARS-CoV-2 in specimens such as nasal or oropharyngeal swabs within 5 days prior to D1 (≤5 days from D1) using nucleic acid amplification assays.
  6. Requirements for laboratory test values, including:

     * Alanine aminotransferase (AST) ≤ 2.5×ULN
     * Aspartate aminotransferase (ALT) ≤ 2.5×ULN
     * Total bilirubin (TBIL) ≤ 2 x ULN (≤ 3.0 x ULN if diagnosed with Gilbert's syndrome)
     * Absolute neutrophil count (ANC) ≥ 1.5×109/L
     * Platelet (PLT)≥ 100 ×109/L
     * Hemoglobin (HB) ≥ 110 g/L
     * International Normalized Ratio (INR) <1.5
     * Partially activated prothrombin time (APTT) < 1.5×ULN
     * Creatinine clearance (according to CKD-EPI formula) ≥ 45mL/min
  7. QTcF ≤ 450msec (male); QTcF ≤ 470msec (female).
  8. Must be willing and able to comply with all planned study procedures.
  9. Women of childbearing potential (WOCBP) (infertile women defined as having undergone hysterectomy or bilateral oophorectomy or bilateral salpingectomy or bilateral tubal ligation/closure, or who are infertile due to a congenital or acquired condition or spontaneously menopausal for ≥ 12 months) must have a negative blood pregnancy test during screening. Fertility female and male subjects must use a highly effective method ofcontraception from the screening period to 90 days after the last dose of study drug.

Exclusion Criteria (applicable to subjects in both parts):

1. Subjects who faint with needles, faint with blood, or have difficulty collecting venous blood.
2. Known hypersensitivity to any of the ingredients of this product.
3. Participated in an interventional clinical trial within 30 days before D1 or within 5 half-lives (whichever is longer).
4. Subjects who have a history of gastrointestinal (such as duodenal ulcer, gastrointestinal bleeding), liver or kidney-related medical history, or other medical history that may affect the absorption, distribution, metabolism, and excretion of oral drugs as assessed by the investigator.
5. Subjects who have undergone major surgery within 3 months prior to screening, or who have not fully recovered from surgery, or who plan to undergo surgery during the study period.
6. Take foods, juices or beverages containing alcohol, grapefruit, lime, cinchona bark and quinine within 24 hours prior to D1.
7. Use of BCRP substrate drugs within 7 days prior to D1 (see "6.5.1 Prohibited Drugs and Treatments").
8. History of substance abuse within 2 years prior to screening.
9. Subjects who have donated blood (including blood components donation) or lost more than 400 mL of blood within 3 months prior to screening.
10. History of alcohol abuse (defined as: more than 14 units of alcohol per week, 1 unit = 150 mL of wine, 360 mL of beer, or 45 mL of spirit containing 40% alcohol) within 3 months prior to screening.
11. Refusal to abstain from smoking after signing the informed consent form and during the study.
12. Excessive consumption of tea, coffee or caffeinated beverages (defined as: at least 8 cups per day, 1 cup = 250 ml) within 3 months prior to screening.
13. Currently pregnant or breastfeeding.
14. According to the investigator's judgment, the subject has any other disease or condition that may affect the normal completion of the study or the evaluation of the study data, or other conditions that are not suitable for participation in this study.

    * Healthy subjects are not allowed to join the part 1 if they meet any of the following criteria:

      1. Relevant history or clinical signs or symptoms associated with clinically significant diseases of the metabolic/endocrine system, heart, liver, kidney, hematolymphatic system, respiratory system, immune system, digestive system, genitourinary system, neurological or psychiatric system within 3 months prior to and during the screening period as assessed by the investigator.
      2. History of fever within 14 days prior to D1.
      3. Liver function test indicators meet the following requirements, including:

         * Alanine aminotransferase (AST) > 1.5 x ULN, or
         * Aspartate aminotransferase (ALT) > 1.5×ULN
      4. QTcF > 450msec (male); QTcF > 470msec (female).
      5. Take any over-the-counter drugs (including but not limited to vitamins, prophylaxis, botanical health products, etc.) or any prescription drugs within 14 days prior to D1 or within 5 half-lives (whichever is longer) (see Exclusion Criteria 13 for BCRP substrate drug limitations) and Chinese herbal medicines, excluding contraceptive drugs or topical drugs that can be applied according to the investigator's assessment.
      6. Subjects who have been vaccinated within 14 days prior to D1, or who plan to be vaccinated during the study.
      7. Positive test for hepatitis B surface antigen (HBsAg), hepatitis C virus (HCV) antibody, and human immunodeficiency virus (HIV) antibody.
      8. On D-1, the nucleic acid amplification detection method will be used to test positive for SARS-CoV-2 in specimens such as nasal or oropharyngeal swabs.
    * SARS-CoV-2 positive subjects are not allowed to join the part 2 if they meet any of the following criteria:

      1. History of COVID-19-related hospitalization within 3 months prior to D1.
      2. According to the investigator's judgment, the subject may progress to severe/critical COVID-19 before randomization.
      3. Within 24 hours prior to D1 (≤24h from D1), SpO2 ≤ 93% or PaO2/FiO2 ≤300 in indoor air at sea level, or respiratory rate ≥30 times/min, or heart rate ≥125 times/min.
      4. Requires mechanical ventilation or anticipates an urgent need for mechanical ventilation.
      5. Suspected or diagnosed serious bacterial, fungal, viral, or other infection (except for COVID-19 infection), or would affect the endpoint assessment of this study according to the investigator assessment.
      6. Active or uncontrolled liver disease: including primary biliary cirrhosis, Child-Pugh class B or C, acute liver failure, etc.
      7. Being on dialysis.
      8. Use any drug known to strongly induce or strongly inhibit CYP3A4 enzyme metabolism within 7 days prior to D1 .
      9. Treatment of COVID-19 with systemic or inhaled steroids within 30 days prior to D1 (long-term stable dose therapy for chronic concomitant disease, without increasing dose).
      10. Have previously received COVID-19 patients' convalescent plasma or anti-SARS-CoV-2 neutralizing antibody or related antiviral therapy.
      11. Subjects who have been vaccinated within 14 days prior to D1, or who plan to be vaccinated during the study.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 79 (Actual)
Dates: Start 2022-09-16 (Actual); Primary Completion 2022-12-21 (Actual); Study Completion 2023-03-29 (Actual)

PRIMARY OUTCOMES:
AE, laboratory tests, thyroid function, physical examination, vital signs. | Day 7 for part 1 and day 29 for part 2.
  Incidence and severity of AEs up to 6 days for part 1 and 21 days for part 2 post-dosing.

SECONDARY OUTCOMES:
Proportion of changes from baseline in SARS-CoV-2 RNA quantification levels on D3, D5, D7, D10, D14, D21, D29. | Day3, Day5, Day7, Day10, Day14, Day21, Day29
  2 nasal swabs will be taken from both nostrils for RNA test
Proportion of SARS-CoV-2 RNA quantification levels below the lower limit of quantification on D3, D5, D7, D10, D14, D21, D29. | Day3, Day5, Day7, Day10, Day14, Day21, Day29.
  2 nasal swabs will be taken from both nostrils for RNA test
Pharmacokinetic parameter of AUC | Day1, Day2, Day3 for part 1 and Day1, Day6, Day7, Day8 for part 2
  Area under the concentration-time curve from time 0 to Day1, Day2, Day3 for part 1 and Day1, Day6, Day7, Day8 for part 2
Pharmacokinetic parameter of Cmax | Day1, Day2, Day3 for part 1 and Day1, Day6, Day7, Day8 for part 2
  Measured by maximum observed concentration
Pharmacokinetic parameter of Tmax | Day1, Day2, Day3 for part 1 and Day1, Day6, Day7, Day8 for part 2
  Measured by time to maximum observed concentration
Pharmacokinetic parameter of t½ | Day1, Day2, Day3 for part 1 and Day1, Day6, Day7, Day8 for part 2
  Terminal elimination half-life after dosing

CONTACTS AND LOCATIONS:
Locations (1):
- The Third People's Hospital Of Shenzhen, Shenzhen, Guangdong, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Mao L, Shaabani N, Zhang X, Jin C, Xu W, Argent C, Kushnareva Y, Powers C, Stegman K, Liu J, Xie H, Xu C, Bao Y, Xu L, Zhang Y, Yang H, Qian S, Hu Y, Shao J, Zhang C, Li T, Li Y, Liu N, Lin Z, Wang S, Wang C, Shen W, Lin Y, Shu D, Zhu Z, Kotoi O, Kerwin L, Han Q, Chumakova L, Teijaro J, Royal M, Brunswick M, Allen R, Ji H, Lu H, Xu X. Olgotrelvir, a dual inhibitor of SARS-CoV-2 Mpro and cathepsin L, as a standalone antiviral oral intervention candidate for COVID-19. Med. 2024 Jan 12;5(1):42-61.e23. doi: 10.1016/j.medj.2023.12.004. Epub 2024 Jan 4. PMID 38181791